CLINICAL TRIAL: NCT01855308
Title: Single Site Robotic Cholecystectomy in Non Selected Patients
Acronym: SSRC
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 307021; 307021 (Other: UC Davis)
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single site robotic chole: Cholecystectomy performed through a single incision with the robot.
  Interventions: Procedure: Single site robotic chole; Device: da Vinci Si Surgical System

INTERVENTIONS:
Procedure: Single site robotic chole — Cholecystectomy
Device: da Vinci Si Surgical System — minimally invasive robotic surgical system designed to facilitate complex procedures

SUMMARY:
This is a study of new technology to allow gallbladder removal through a single small surgical incision. A surgical robot is utilized to help navigate the small space. In this study, patient characteristics are broad to assess how applicable the procedure is to everyone.

ELIGIBILITY:
Inclusion Criteria:

* presence of symptomatic gallstones

Exclusion Criteria:

* significant previous open abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are referred to the surgery program with non-emergency gallbladder disease, for which cholecystectomy is indicated, will be given the opportunity to participate. Referred patients typically come from the primary care setting. The demographic composition of the study population will depend in the patient referred to the program.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Completion of procedure by SSRC | At time of surgery

SECONDARY OUTCOMES:
Adverse events to study participants (e.g. bile duct injury, hemorrhage) | At time of procedure and in clinic up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Ali, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States